CLINICAL TRIAL: NCT07288944
Title: A Comparison of Two Phosphate Replacement Protocols for Critically Ill Patients Treated in an Intensive Care Unit: a Cluster, Crossover, Comparative Effectiveness, Randomised, Controlled Trial
Brief Title: Protocolised Management of Phosphate Replacement Trial
Acronym: PROMPT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Caboolture Hospital (Other Government)
Collaborators: Queensland University of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HREC/2025/MNH/121108
Record Dates: First submitted 2025-11-20; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Phosphate Deficiency; Hypophosphatemia; Protocol Optimization; Critical Care, Intensive Care
Keywords: Phosphate Protocol; Critical Care; Intensive Care; Hypophosphatemia; Phosphate Deficiency
MeSH Terms: conditions — Hypophosphatemia

STUDY DESIGN:
Intervention Model Description: A cluster, crossover, electronic medical record (EMR)-integrated, randomised, controlled trial (RCT) that will compare liberal versus restrictive protocolised replacement of phosphate in critically ill patients admitted to intensive care units (ICU).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liberal Phosphate Replacement Protocol (Active Comparator): The liberal group, a recommendation for phosphate replacement would be given if the serum phosphate concentration was 0.79 mmol/L, but not if 0.80 mmol/L.
  Interventions: Other: Liberal Phosphate Replacement Protocol
- Conservative Phosphate Replacement Protocol (Active Comparator): The restrictive protocol will recommend phosphate replacement to commence at a threshold of 0.50 mmol/L, and the liberal protocol at 0.80 mmol/L.
  Interventions: Other: Restrictive Phosphate Replacement Protocol

INTERVENTIONS:
Other: Liberal Phosphate Replacement Protocol — The liberal group, a recommendation for phosphate replacement would be given if the serum phosphate concentration was 0.79 mmol/L, but not if 0.80 mmol/L.
  Arms: Liberal Phosphate Replacement Protocol
Other: Restrictive Phosphate Replacement Protocol — The restrictive protocol will recommend phosphate replacement to commence at a threshold of 0.50 mmol/L, and the liberal protocol at 0.80 mmol/L.
  Arms: Conservative Phosphate Replacement Protocol

SUMMARY:
The aim of this cluster, crossover, randomised controlled trial is to compare two standard arms of treatment for the replacement of phosphate in critically ill patients.

We hypothesise that protocolised restricted phosphate replacement, compared to protocolised liberal phosphate replacement, will result in reduced administration of phosphate with similar clinical outcomes.

All eligible Intensive Care Unit (ICU) patients will be included during their admission with the selected protocol for that period as per usual practice and treatment standards.

DETAILED DESCRIPTION:
This study looks to compare liberal and restrictive phosphate replacement protocols (each arm is a current "standard of care" already used in practice) to investigate whether restrictive phosphate replacement in critically ill patients leads to reduced phosphate administration and/or equivalent patient outcomes.

Derangements of serum phosphate concentrations are common among ICU patients; high and low levels variably associated with worse outcomes. The PROMPT trial will compare two standard arms of treatment for the replacement of phosphate in critically ill patients. Phosphate is currently replaced routinely in ICU's however there is not a standardised evidence-based guideline to effectively guide phosphate administration for ICU patients

This is a cluster, crossover, electronic medical record integrated, randomised, controlled trial. Sites (not patients) will be randomised to wither the liberal or restrictive phosphate replacement protocol for a 6-month period, followed by a 1-month washout period, before switching to the next protocol for the preceding 6-month period. The allocated phosphate replacement protocol will be updated in the electronic medical record to be followed; this process is already part of normal clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients admitted to participating intensive care units during the study period.

Exclusion Criteria:

* There will be no specific exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
non-inferiority for days alive and free of the intensive care unit (ICU) up to 30 days (DAF-ICU-30) | 30 Days post study enrolment
  The primary outcome will be assessed as non-inferiority in the number of days alive and free of ICU within 30 days from study enrolment. ICU length of stay will be used to calculate. This measure is reported on a continuous scale ranging from 0 (worst outcome: death or full ICU stay) to 30 (best outcome: alive and ICU-free for all 30 days), where higher scores indicate a better outcome. The difference between groups will be expressed as a mean difference with 95% confidence intervals.

SECONDARY OUTCOMES:
Phosphate usage | individual arm and total quantities used over 12-month study period
  Quantities of intravenous and oral phosphate replaced (total and individually)
Patients receiving phosphate | total proportion of patients receiving phosphate throughout 12-month study period
  Proportion of patients receiving any phosphate replacement
Hospital Length of Stay | hospital admission to hospital discharge throughout 12-month study period
  Total time spent in hospital - hospital admission time to hospital discharge time
Hospital Mortality | hospital admission to hospital discharge throughout 12-month study period
  hospital mortality rates for all participants throughout study period
cardiac rhythm disturbance | ICU admission to ICU discharge, throughout 12-month study period
  Symptomatic cardiac rhythm disturbance (cardiac arrhythmia that requires treatment with chemical or electric cardioversion)
Mechanical ventilation hours | hospital admission to hospital discharge, throughout 12-month study period
  Hours of invasive mechanical ventilation
Tracheal reintubation | hospital admission to hospital discharge, throughout 12-month study period
  Tracheal intubation requirement during admission

CONTACTS AND LOCATIONS:
Overall Officials: Mahesh Ramanan, Principal Investigator — +61 7 5433 8888

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramanan M, Tabah A, Affleck J, Edwards F, White KC, Attokaran A, Laupland K. Hypophosphataemia in Critical Illness: A Narrative Review. J Clin Med. 2024 Nov 26;13(23):7165. doi: 10.3390/jcm13237165. PMID 39685625
- [Background] Sin JCK, Laupland KB, Ramanan M, Tabah A. Phosphate abnormalities and outcomes among admissions to the intensive care unit: A retrospective multicentre cohort study. J Crit Care. 2021 Aug;64:154-159. doi: 10.1016/j.jcrc.2021.03.012. Epub 2021 Apr 18. PMID 33906104